CLINICAL TRIAL: NCT05232552
Title: Safety and Efficacy of Anlotinib With Chemoradiation for Patients With Locally Advanced Nasopharyngeal Carcinoma: a Phase 2 Study
Brief Title: Study of Anlotinib With Chemoradiation for Patients With Locally Advanced Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Chen Xiaozhong, Director, Head of Radiation department, Principal Investigator, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-anlotinib 1
Record Dates: First submitted 2021-05-23; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2021-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib (Experimental): 3 cycles of anlotinib (12mg, d1-14)was given concurrently with docetaxel plus cisplatin chemotherapy as induction , then 2 additional cycles of anlotinib concurrent with definitive chemoradiation (IMRT with conccurent cisplatin)
  Interventions: Drug: Anlotinib hydrochloride; Drug: induction chemotherapy; Radiation: concurrent chemoradiation

INTERVENTIONS:
Drug: Anlotinib hydrochloride — anlotinib was administered orally 12mg daily for 14 days concurrent with inductive chemotherapy (TP ) for 3 cycles and definitive chemoradiation for additional 2 cycles
Drug: induction chemotherapy — docetaxel 75mg/m2 d1 plus DDP 75mg/m2 d1 for 3 cycles every 21days
  Other Names: IC
Radiation: concurrent chemoradiation — definitive IMRT (GTV>66Gy) concurrent with 2 cycles of DDP (100mg/m2 d1) and anlotinib (12mg d1-14) every 21 days
  Other Names: CCRT

SUMMARY:
anlotinib was added to TP inductive chemotherapy and definitive chemoradiation in nasopharyngeal carcinoma patients with N2-3 disease with necrosis or/and ECM

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed nasopharyngeal carcinoma confirmed by histology/cytology ;
2. N2-3 disease (UICC/AJCC 8th) with necrosis or/and ECM;
3. with sufficient organ and bone marrow function;
4. ECOG (Eastern US Cooperative Oncology Group) score < 3
5. with good compliance and cooperation to treatment and follow-up
6. agree to use effective methods of contraception during the study period and within 180 days of the last study administration.

Exclusion Criteria:

1. patients with other malignant tumors diagnosed within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) ) And T1 (tumor infiltration basement membrane)]
2. patients with bleeding events NCI-CTC AE V5.0 grade ≥ 3, unhealed wounds, ulcers or fracture;
3. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS), active hepatitis B (HBV DNA ≥ 500 IU / ml), hepatitis C (HCV antibody positive, and HCV RNA higher than the detection limit of the analysis method) or co infection with hepatitis B and C.
4. Active infection (e.g. intravenous drip of antibiotics, antifungal or antiviral drugs) or fever of unknown origin >38.5℃ 1 weeks ago (except for tumor related fever determined by researchers).
5. Abnormal coagulation (INR > 1.5 or APTT > 1.5 × ULN), bleeding tendency or undergoing thrombolysis or anticoagulation. Long term anticoagulation with warfarin or heparin or long-term antiplatelet therapy is required.
6. serious physical or mental illness or laboratory abnormalities may increase the risk of participating in the study
7. Allergy to the drugs in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | induction phase ; 3 months after chemoradiation
  tumor objective response rate

SECONDARY OUTCOMES:
PFS | 3year
  progression-free survival
LRR | 3 years
  local relapse rate
RRR | 3 years
  regional relapse rate

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
IPD could be shared with reasonable reasons